CLINICAL TRIAL: NCT04998604
Title: A Randomized, Double-blind, Head-to-head Comparison of Dupilumab Versus Omalizumab in Severe Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) and Comorbid Asthma Patients
Brief Title: EValuating trEatment RESponses of Dupilumab Versus Omalizumab in Type 2 Patients
Acronym: EVEREST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPS16747; U1111-1255-4713 (Registry Identifier: ICTRP); 2021-000829-27 (EudraCT Number)
Record Dates: First submitted 2021-08-09; First posted 2021-08-10 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo injections will be administered as needed to blind the number of active dupilumab and omalizumab injections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab 300 mg Q2W (Experimental): Participants received dupilumab 300 milligrams (mg) subcutaneous (SC) injection every 2 weeks (Q2W) for 24 weeks.
  Interventions: Drug: Dupilumab; Drug: Placebo
- Omalizumab 75 to 600 mg Q2W/Q4W (Experimental): Participants received omalizumab 75 to 600 mg SC injection Q2W/every 4 weeks (Q4W) based on their serum immunoglobulin E (IgE) levels and body weight for 24 weeks.
  Interventions: Drug: Omalizumab; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — solution for injection subcutaneous
  Other Names: SAR231893 Dupixent
  Arms: Dupilumab 300 mg Q2W
Drug: Omalizumab — solution for injection subcutaneous
  Other Names: Xolair
  Arms: Omalizumab 75 to 600 mg Q2W/Q4W
Drug: Placebo — solution for injection subcutaneous

SUMMARY:
Primary Objective

-To evaluate the efficacy of dupilumab compared to omalizumab in reducing the polyp size and improving sense of smell

Secondary Objectives

* To evaluate the efficacy of dupilumab in improving chronic rhinosinusitis with nasal polyps (CRSwNP) symptoms at Week 24 compared to omalizumab
* To evaluate the efficacy of dupilumab in improving CRSwNP total symptom score (TSS) at Week 24 compared to omalizumab
* To evaluate the effect of dupilumab on health related quality of life (HRQoL) at week 24 compared to omalizumab
* To evaluate the efficacy of dupilumab in improving nasal peak inspiratory flow at Week 24 compared to omalizumab
* To evaluate the effect of dupilumab on CRSwNP overall disease severity at Week 24 compared to omalizumab
* To evaluate the safety of dupilumab and omalizumab

DETAILED DESCRIPTION:
Study duration per participant will be 38 weeks. The study will comprise 3 periods: 28 days ± 3 days screening and run-in period; 24 weeks Randomized investigational medicinal product (IMP) intervention period; up to 12 weeks follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 (or the legal age of consent in the jurisdiction in which the study is taking place) years of age inclusive, at the time of signing the informed consent.
* Participants with bilateral sino-nasal polyposis, that despite prior treatment with Systemic corticosteroids (SCS) anytime within the past 2 years; and/or medical contraindication/intolerance to SCS; and/or prior surgery for NP have:

  * An endoscopic bilateral NPS of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity) at visit 1; AND
  * Ongoing symptoms of Nasal congestion/blockade/obstruction and loss of smell for at least 8 weeks before screening (Visit 1), AND
  * Nasal congestion/blockade/obstruction and a weekly average severity greater than 1 in the 7 days before randomization (Visit 2) AND
  * loss of smell symptom severity score 2 or 3 at screening (Visit 1) and a weekly average severity of greater than 1 in the 7 days before randomization (Visit 2).
* Participants with a physician diagnosis of asthma based on the Global Initiative for Asthma (GINA) 2020 treated with low, medium or high dose inhaled corticosteroids (ICS) and a second controller (ie, LABA), a third controller is allowed but not mandatory. The dose regimen was to be stable for at least 1 month before Visit 1 (screening visit) and during the screening and run-in period.
* Asthma Control Questionnaire 5-question version (ACQ-5) score ≥1.5 at Visits 1 or 2.
* Treatment with intranasal mometasone ≥200 μg once daily (QD) (or equivalent of another INCS) for 1 month prior to Visit 1 and during the run-in period (for CRSwNP).
* Eligibility as per omalizumab drug-dosing table (serum IgE level ≥30 to ≤1500 IU/mL and body weight ≥30 to ≤150 kg) and ability to be dosed per the dosing table.

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria apply:

* Participants who underwent any sinus intranasal surgery (including polypectomy) within 6 months before Visit 1.
* Participants who had a sino-nasal surgery changing the lateral wall structure of the nose, making impossible the evaluation of NPS.
* Participants with conditions/concomitant diseases making them non evaluable at Visit 1 or for the primary efficacy endpoint such as: Antrochoanal polyps, Nasal septal deviation that would occlude at least one nostril, Acute sinusitis, nasal infection, or upper respiratory infection.
* Severe asthma exacerbation requiring treatment with SCS in the last 4 weeks prior to Visit 1 and during screening.
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study
* Diagnosed with, suspected of, or at high risk of endoparasitic infection, and/or use of antiparasitic drugs within 2 weeks before Visit 1 (screening visit) or during the screening and run-in period.
* History of human immunodeficiency virus (HIV) infection or positive HIV 1/2 serology at Visit 1 (screening visit).
* Known or suspected immunodeficiency, including history of invasive opportunistic infections
* Active malignancy or history of malignancy within 5 years before Visit 1 (screening visit), except completely treated in situ carcinoma of the cervix and completely treated and resolved non metastatic squamous or basal cell carcinoma of the skin.
* History of systemic hypersensitivity or anaphylaxis to dupilumab and omalizumab, including any excipient
* Treatment with a live (attenuated) vaccine within 4 weeks before Visit 1 (screening visit).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (87):
- United States (16):
  - Cedars Sinai Medical Center Site Number : 8400026, Los Angeles, California
  - Asthma Allergy & Immunology Clinical Research Unit Site Number : 8400027, Tampa, Florida
  - Northwestern University Site Number : 8400001, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advanced ENT and Allergy Site Number : 8400013, Louisville, Kentucky
  - University of Missouri Health Care - University Hospital Site Number : 8400016, Columbia, Missouri
  - Northwell Health Site Number : 8400044, Great Neck, New York
  - University of Rochester Site Number : 8400015, Rochester, New York
  - Cleveland Clinic Foundation Site Number : 8400029, Cleveland, Ohio
  - Optimed Research, LTD Site Number : 8400014, Columbus, Ohio
  - Allergy, Asthma and Clinical Research Center Site Number : 8400037, Oklahoma City, Oklahoma
  - Essential Medical Research, LLC Site Number : 8400024, Tulsa, Oklahoma
  - Oregon Health & Science University Site Number : 8400031, Portland, Oregon
  - University of Texas Health Science Center- Site Number : 8400019, Houston, Texas
  - Chryaslis Clinical Research Site Number : 8400017, St. George, Utah
  - Eastern Virginia Medical School Site Number : 8400010, Norfolk, Virginia
- Belgium (3):
  - Investigational Site Number : 0560001, Ghent
  - Investigational Site Number : 0560002, Leuven
  - Investigational Site Number : 0560003, Woluwe-Saint-Lambert
- Canada (3):
  - Investigational Site Number : 1240004, London, Ontario
  - Investigational Site Number : 1240002, Montreal, Quebec
  - Investigational Site Number : 1240003, Québec
- Czechia (9):
  - Investigational Site Number : 2030007, Benešov
  - Investigational Site Number : 2030001, Hradec Králové
  - Investigational Site Number : 2030003, Ostrava - Poruba
  - Investigational Site Number : 2030002, Pardubice
  - Investigational Site Number : 2030012, Pilsen
  - Investigational Site Number : 2030010, Prague
  - Investigational Site Number : 2030006, Prague
  - Investigational Site Number : 2030008, Prague
  - Investigational Site Number : 2030004, Praha 5 - Motole
- Denmark (2):
  - Investigational Site Number : 2080003, Aarhus
  - Investigational Site Number : 2080001, Copenhagen
- Finland (2):
  - Investigational Site Number : 2460003, Helsinki
  - Investigational Site Number : 2460002, Tampere
- France (7):
  - Investigational Site Number : 2500009, Créteil
  - Investigational Site Number : 2500006, La Roche-sur-Yon
  - Investigational Site Number : 2500008, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500002, Lille
  - Investigational Site Number : 2500004, Marseille
  - Investigational Site Number : 2500005, Montpellier
  - Investigational Site Number : 2500007, Toulouse
- Germany (4):
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760004, Düsseldorf
  - Investigational Site Number : 2760003, München
  - Investigational Site Number : 2760001, Münster
- Hungary (6):
  - Investigational Site Number : 3480007, Budapest
  - Investigational Site Number : 3480004, Budapest
  - Investigational Site Number : 3480005, Debrecen
  - Investigational Site Number : 3480006, Edelény
  - Investigational Site Number : 3480002, Pécs
  - Investigational Site Number : 3480001, Szeged
- Italy (6):
  - Investigational Site Number : 3800002, Rome, Lazio
  - Investigational Site Number : 3800001, Rozzano, Lombardy
  - Investigational Site Number : 3800003, Catania
  - Investigational Site Number : 3800004, Florence
  - Investigational Site Number : 3800006, Milan
  - Investigational Site Number : 3800005, Varese
- Mexico (3):
  - Investigational Site Number : 4840003, Guadalajara, Jalisco
  - Investigational Site Number : 4840002, Chihuahua City
  - Investigational Site Number : 4840004, Durango
- Poland (6):
  - Investigational Site Number : 6160004, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160008, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160005, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160001, Krakow
  - Investigational Site Number : 6160007, Lodz
  - Investigational Site Number : 6160006, Środa Wielkopolska
- Portugal (5):
  - Investigational Site Number : 6200005, Almada
  - Investigational Site Number : 6200003, Aveiro
  - Investigational Site Number : 6200006, Guimarães
  - Investigational Site Number : 6200001, Matosinhos Municipality
  - Investigational Site Number : 6200007, Santa Maria da Feira
- Romania (2):
  - Investigational Site Number : 6420002, Brasov
  - Investigational Site Number : 6420004, Craiova
- Spain (7):
  - Investigational Site Number : 7240001, Seville, Andalusia
  - Investigational Site Number : 7240005, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240008, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Jerez de la Frontera, Cádiz
  - Investigational Site Number : 7240007, Majadahonda, Madrid
  - Investigational Site Number : 7240004, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240006, Pamplona, Navarre
- Sweden (3):
  - Investigational Site Number : 7520003, Gothenburg
  - Investigational Site Number : 7520002, Lund
  - Investigational Site Number : 7520001, Stockholm
- United Kingdom (3):
  - Investigational Site Number : 8260003, Wigan, Lancashire
  - Investigational Site Number : 8260002, Manchester
  - Investigational Site Number : 8260001, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] De Corso E, Canonica GW, Heffler E, Springer M, Grzegorzek T, Viana M, Horvath Z, Mullol J, Gevaert P, Michel J, Peters AT, Wagenmann M, Zaghloul S, Zhang M, Corbett M, Nash S, Angello JT, Radwan A, Deniz Y, Martin A, Hellings PW. Dupilumab versus omalizumab in patients with chronic rhinosinusitis with nasal polyps and coexisting asthma (EVEREST): a multicentre, randomised, double-blind, head-to-head phase 4 trial. Lancet Respir Med. 2025 Dec;13(12):1067-1077. doi: 10.1016/S2213-2600(25)00287-5. Epub 2025 Sep 28. PMID 41033334
- [Derived] De Prado Gomez PharmD MSc L, Khan Mbbs Mph AH, Peters Md AT, Bachert Md PhD C, Wagenmann Md M, Heffler Md PhD E, Hopkins BMBCh C, Hellings Md PhD PW, Zhang PhD M, Xing PhD J, Rowe Md P, Jacob-Nara Md Mph DHSc JA. Efficacy and Safety of Dupilumab Versus Omalizumab in Chronic Rhinosinusitis With Nasal Polyps and Asthma: EVEREST Trial Design. Am J Rhinol Allergy. 2022 Nov;36(6):788-795. doi: 10.1177/19458924221112211. Epub 2022 Jul 15. PMID 35837739
- See also: LPS16747 Chronic Rhinosinusitis with Nasal Polyps Dupilumab Trial website — https://www.sanofistudies.com/1GHY/
- See also: LPS16747 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25289&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 87 active centers in 17 countries. A total of 819 participants were screened between 27 September 2021 and 25 April 2024, of which 459 participants were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 360 participants were randomized in a 1:1 ratio to receive either dupilumab or omalizumab in the study. Randomization was stratified by prior surgery for nasal polyp, inhaled corticosteroids (ICS) doses (low versus medium/high dose ICS), presence of aspirin-exacerbated respiratory disease (AERD) and region [Eastern European (EE) versus Rest of the World (ROW)].
Period: Overall Study
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Started | 181 | 179
Randomized and Treated | 179 | 173
Completed | 174 | 165
Not Completed | 7 | 14
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Not related to coronavirus disease 2019 pandemic | 2 | 8

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Dupilumab 300 mg Q2W: Participants received dupilumab 300 mg SC injection Q2W for 24 weeks.
- Omalizumab 75 to 600 mg Q2W/Q4W: Participants received omalizumab 75 to 600 mg SC injection Q2W/Q4W based on their serum IgE levels and body weight for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W | Total
Number analyzed (Participants) | 181 | 179 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.33) | 52.1 (12.90) | 51.5 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 88 | 162
  Male | 107 | 91 | 198
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Black or African American | 2 | 1 | 3
  White | 171 | 170 | 341
  Multiple | 0 | 1 | 1
  Not Reported | 6 | 2 | 8
  Unknown | 1 | 2 | 3
Nasal Polyp Score (NPS) [Mean (Standard Deviation); unit: score on a scale] — The NPS was assessed by the independent physician to grade the extent/severity of nasal polyps based on evaluation by nasal endoscopy. The NPS scores for each nostril was graded based on polyp size from 0 (no polyps) to 4 (large polyps causing complete obstruction of the inferior nasal cavity). The total NPS score was calculated as the sum of right and left nostril scores and ranged from 0 (no polyps) to 8 (large polyps). Higher scores indicated more extensive or severe nasal polyps.
  score on a scale | 6.11 (1.165) | 6.15 (1.277) | 6.13 (1.220)
University of Pennsylvania Smell Identification Test (UPSIT) [Mean (Standard Deviation); unit: score on a scale] — The UPSIT was a 40-item test to quantitatively assess human olfactory function. The UPSIT test consisted of 4 booklets, each containing 10 odorants with 1 odorant per page. The participant was asked to release the odorant by rubbing the brown-strip (contained odorant microcapsules) with the tip of a pencil and to indicate which of 4 words best described the odor. Thus, each participant received a score out of 40 possible correct answers. The total UPSIT score ranged from 0 (loss of smell/anosmia) to 40 (normal sense of smell/normosmia). Higher scores indicated better olfactory function. Population: Only number of participants evaluable for the specified baseline measure are reported.
  score on a scale
    number analyzed (Participants) | 180 | 175 | 355
    (all) | 11.1 (5.45) | 11.0 (6.13) | 11.1 (5.79)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Nasal Polyp Score
Description: The NPS was assessed by the independent physician to grade the extent/severity of nasal polyps based on evaluation by nasal endoscopy. The NPS scores for each nostril was graded based on polyp size from 0 (no polyps) to 4 (large polyps causing complete obstruction of the inferior nasal cavity). The total NPS score was calculated as the sum of right and left nostril scores and ranged from 0 (no polyps) to 8 (large polyps). Higher scores indicated more extensive or severe nasal polyps. Negative change from baseline indicated less severity of nasal polyps. Baseline was defined as the last available valid (non-missing) value up to and including the day of first administration of study treatment.
Time Frame: Baseline (Day 1) and Week 24
Population: The ITT analysis set included all randomized participants. Only participants with data collected at Week 24 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 172 | 165
score on a scale | -2.65 [-2.95 to -2.36] | -1.05 [-1.35 to -0.75]
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Omalizumab 75 to 600 mg Q2W/Q4W; A hierarchical testing procedure was used to control the type-I error and handle multiple secondary endpoint analysis. Testing was performed sequentially in order the endpoints were reported and continued when primary endpoint was statistically significant at 2-sided 0.05; Test type: Superiority — At each post-baseline visit, each of the imputed complete data was analyzed by fitting an analysis of covariance (ANCOVA) model with the corresponding baseline value, study treatment (dupilumab, omalizumab), prior surgery (yes, no), ICS doses (low, medium/high), presence of AERD (yes, no), region (EE, ROW) as covariates; p < 0.001, ANCOVA — The threshold for statistical significance was 0.05 level; Least squares (LS) mean difference = -1.60, 95% CI 2-sided [-1.96 to -1.25], Standard Error of Mean 0.182

2. Primary Outcome: Change From Baseline to Week 24 in University of Pennsylvania Smell Identification Test
Description: The UPSIT was a 40-item test to quantitatively assess human olfactory function. The UPSIT test consisted of 4 booklets, each containing 10 odorants with 1 odorant per page. The participant was asked to release the odorant by rubbing the brown-strip (contained odorant microcapsules) with the tip of a pencil and to indicate which of 4 words best described the odor. Thus, each participant received a score out of 40 possible correct answers. The total UPSIT score ranged from 0 (loss of smell/anosmia) to 40 (normal sense of smell/normosmia). Higher scores indicated better olfactory function. Positive change from baseline indicated normal olfactory function. Baseline was defined as the last available valid (non-missing) value up to and including the day of first administration of study treatment.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 173 | 166
score on a scale | 12.7 [11.3 to 14.1] | 4.7 [3.2 to 6.1]
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Omalizumab 75 to 600 mg Q2W/Q4W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority — At each post-baseline visit, each of the imputed complete data was analyzed by fitting an ANCOVA model with the corresponding baseline value, study treatment (dupilumab, omalizumab), prior surgery (yes, no), ICS doses (low, medium/high), presence of AERD (yes, no), region (EE, ROW) as covariates; p < 0.001, ANCOVA — The threshold for statistical significance was 0.05 level; LS mean difference = 8.0, 95% CI 2-sided [6.3 to 9.7], Standard Error of Mean 0.88

3. Secondary Outcome: Change From Baseline to Week 24 in the Loss of Smell Score of the Chronic Rhinosinusitis With Nasal Polyp (CRSwNP) Nasal Symptom Diary
Description: The nasal symptom diary was designed to assess the severity of chronic rhinosinusitis nasal symptoms daily. These symptoms included nasal congestion (NC)/obstruction, loss of smell, anterior rhinorrhea, and posterior rhinorrhea. The severity of loss of smell was scored by participants using a scale ranged from 0 to 3 (where, 0= no symptoms, 1= mild symptoms, 2= moderate symptoms and 3= severe symptoms that were hard to tolerate, caused interference with activities, or daily living). Higher scores indicated greater symptom severity. Negative change from baseline indicated less severe symptom. Baseline value was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (average of Day -6 to Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 170 | 164
score on a scale | -1.55 [-1.71 to -1.38] | -0.74 [-0.90 to -0.57]
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Omalizumab 75 to 600 mg Q2W/Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Each of the imputed complete data was analyzed by fitting an ANCOVA model with the corresponding baseline value, study treatment (dupilumab, omalizumab), prior surgery (yes, no), ICS doses (low, medium/high), presence of AERD (yes, no), region (EE, ROW) as covariates; p < 0.001, ANCOVA — The threshold for statistical significance was 0.05 level; LS mean difference = -0.81, 95% CI 2-sided [-1.01 to -0.61], Standard Error of Mean 0.101

4. Secondary Outcome: Change From Baseline to Week 24 in the Nasal Congestion Score of the Chronic Rhinosinusitis With Nasal Polyp Nasal Symptom Diary
Description: The nasal symptom diary was designed to assess the severity of chronic rhinosinusitis nasal symptoms daily. These symptoms included NC/obstruction, loss of smell, anterior rhinorrhea, and posterior rhinorrhea. The severity of NC was scored by participants using a scale ranged from 0 to 3 (where, 0= no symptoms, 1= mild symptoms, 2= moderate symptoms and 3= severe symptoms that were hard to tolerate, caused interference with activities, or daily living). Higher scores indicated greater symptom severity. Negative change from baseline indicated less severe symptom. Baseline value was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (average of Day -6 to Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 170 | 164
score on a scale | -1.63 [-1.76 to -1.49] | -1.05 [-1.18 to -0.91]
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Omalizumab 75 to 600 mg Q2W/Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA — The threshold for statistical significance was 0.05 level; LS mean difference = -0.58, 95% CI 2-sided [-0.74 to -0.42], Standard Error of Mean 0.082

5. Secondary Outcome: Change From Baseline to Week 24 in Total Symptom Score (TSS) Derived From the Chronic Rhinosinusitis With Nasal Polyp Nasal Symptom Diary
Description: The TSS is a composite score consisted of the following symptoms assessed daily in the morning: NC/obstruction, decreased/loss of sense of smell, and rhinorrhea (average of anterior/posterior nasal discharge). Each item was scored on a scale ranged from 0 to 3 (where, 0= no symptoms, 1= mild symptoms, 2= moderate symptoms and 3= severe symptoms that were hard to tolerate, and caused interference with activities, or daily living). Higher score indicated greater symptom severity. The TSS score was calculated by summing the individual symptom score and ranged from 0 (no symptoms) to 9 (severe symptoms). Higher scores on the TSS indicated greater symptom severity. Negative change from baseline indicated less severe symptom. Baseline was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (average of Day -6 to Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 170 | 164
score on a scale | -4.48 [-4.82 to -4.14] | -2.73 [-3.09 to -2.38]
Statistical Analysis 1: Comparison: Dupilumab 300 mg Q2W vs Omalizumab 75 to 600 mg Q2W/Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA — The threshold for statistical significance was 0.05 level; LS mean difference = -1.74, 95% CI 2-sided [-2.15 to -1.33], Standard Error of Mean 0.210

6. Secondary Outcome: Change From Baseline to Week 24 in Sino-Nasal Outcome Test 22-Items (SNOT-22) Total Score
Description: The SNOT-22 is a patient-reported outcome questionnaire designed to assess the impact of chronic rhinosinusitis on participants' health-related quality of life. The SNOT-22 consisted of 22 items covering symptoms, social/emotional impact, productivity, and sleep consequences of chronic rhinosinusitis. Each item was rated on a 6-point Likert scale response option, score ranged from 0 (no problem) to 5 (problem as bad as it can be). The SNOT-22 total score was the sum of each item score, and it ranged from 0 (no problem) to 110 (problem as bad as it can be). Higher scores indicated greater rhinosinusitis-related health burden, meaning for this parameter lower score indicated better condition. Negative change from baseline indicated improvement in health-related quality of life. Baseline was defined as the last available valid (non-missing) value up to and including the day of first administration of study treatment.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 161 | 158
score on a scale | -44.6 [-47.9 to -41.3] | -31.9 [-35.2 to -28.5]

7. Secondary Outcome: Change From Baseline to Week 24 in Sino-Nasal Outcome Test 22-Items: Nasal Domain Score
Description: SNOT-22 is a patient-reported outcome questionnaire designed to assess impact of chronic rhinosinusitis on participants' health-related quality of life. SNOT-22 was categorized into 5 domains: Nasal (items 1, 2, 3, 4, 5, 6, 7 and 12); Ear/Facial (items 8, 9, 10 and 11); Sleep (items 13, 14, 15 and 16); Function (items 17, 18 and 19); Emotion (items 20, 21 and 22). Each item of Nasal domain was rated on a 6-point Likert scale ranged from 0 (no problem) to 5 (problem as bad as it can be) with higher score indicated greater rhinosinusitis-related health burden. Total score of Nasal domain was average score of items of nasal domain, and ranged from 0 (no problem) to 5 (problem as bad as it can be), where higher score indicated greater rhinosinusitis-related health burden. Negative change from baseline indicated improvement in health-related quality of life. Baseline was defined as last available valid (non-missing) value up to and including day of first administration of study treatment.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 161 | 158
score on a scale | -2.4 [-2.6 to -2.2] | -1.6 [-1.8 to -1.4]

8. Secondary Outcome: Change From Baseline to Week 24 in Nasal Peak Inspiratory Flow (NPIF)
Description: The NPIF evaluation represented a physiologic measure of the air flow through both nasal cavities during forced inspiration. The NPIF is the best validated technique for the evaluation of nasal flow through the nose. Participants were issued an NPIF meter and were instructed on the use of the device and written instructions on the use of the NPIF meter was provided. Higher NPIF values were indicative of better nasal air flow. Positive change from baseline indicated better nasal air flow. Baseline was the mean measurement recorded for the 7 days (Day -6 to Day 1) prior to first dose of study treatment.
Time Frame: Baseline (average of Day -6 to Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters per minute
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 169 | 163
Liters per minute | 68.96 [60.90 to 77.02] | 37.69 [29.28 to 46.09]

9. Secondary Outcome: Change From Baseline to Week 24 in Rhinosinusitis Visual Analogue Scale (Rhinosinusitis VAS)
Description: The rhinosinusitis severity VAS was used to evaluate the overall severity of the rhinosinusitis. It is a recommended scale to determine the participant's disease severity and to guide the treatment for chronic rhinosinusitis. The participants were asked to answer the following question: "How troublesome are your symptoms of your rhinosinusitis" on a 10-centimeter VAS from 0 (not troublesome) to 10 (worst thinkable troublesome). Higher scores on the VAS score indicated more severe chronic rhinosinusitis. Negative change from baseline indicated less severity of rhinosinusitis. Baseline was defined as the last available valid (non-missing) value up to and including the day of first administration of study treatment.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 161 | 158
units on a scale | -5.43 [-5.96 to -4.90] | -3.56 [-4.11 to -3.01]

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (SAEs) and Treatment-Emergent Adverse Events of Special Interest (AESIs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required. The TEAEs was defined as an AEs that occurred from the first administration of the study treatment (on Day 1) up to 98 days after the last dose of study treatment administration.
Time Frame: From first dose of study treatment administration (Day 1) up to 98 days after the last dose of study treatment administration (considering the maximum duration of treatment exposure) i.e., up to approximately 329 days
Population: The Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
Number analyzed (Participants) | 179 | 173
Participants
  Any TEAE | 115 | 116
  Any Serious TEAE | 3 | 7
  Any Treatment-Emergent AESI | 4 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs) and other AEs were collected from first dose of study treatment administration (Day 1) up to 98 days after the last dose of study treatment administration (considering the maximum duration of treatment exposure) i.e., up to approximately 329 days. All-cause mortality (deaths) were collected from first dose of study treatment (Day 1) up to end of follow-up for death for each participant, i.e., up to approximately 39 months
Description: Analysis was performed on the safety analysis set.
Arm/Group | Dupilumab 300 mg Q2W | Omalizumab 75 to 600 mg Q2W/Q4W
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/173
Serious Adverse Events (participants affected / at risk) | 3/179 | 7/173
Other Adverse Events (participants affected / at risk) | 48/179 | 53/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg Q2W (N=179) | Omalizumab 75 to 600 mg Q2W/Q4W (N=173)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eosinophilic Granulomatosis With Polyangiitis (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium Avium Complex Infection (Infections and infestations) | 1 (1) | 0 (0)
Neuroborreliosis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia Klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Granulomatosis With Polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg Q2W (N=179) | Omalizumab 75 to 600 mg Q2W/Q4W (N=173)
Nasopharyngitis (Infections and infestations) | 21 (25) | 20 (22)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (12) | 8 (8)
Accidental Overdose (Injury, poisoning and procedural complications) | 12 (14) | 21 (24)
Headache (Nervous system disorders) | 10 (12) | 13 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT04998604/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT04998604/SAP_001.pdf